CLINICAL TRIAL: NCT07008040
Title: Assessing the Effect of the Silver Dressing on Surgical Site Infections in Adult Patients Post Cardiac Surgery: a Single Center Randomized Control Trial
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Principal Investigator, Jennifer De Beer, Dr, King Faisal Specialist Hospital & Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RAC2024-14; RAC 2024-14 (Other Grant/Funding Number: KFSHRC-J); Research Ethics Committee (Other: King Faisal Specialist Hospital and Research Center - Jeddah)
Record Dates: First submitted 2025-05-29; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Surgical Site Infection After Major Surgery; Surgical Site Infections
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: control and intervention group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mepilex Border Opsite dressing (Other): Only foam dressing used in this arm
  Interventions: Other: Silver dressing

INTERVENTIONS:
Other: Silver dressing — Silver dressing will be applied to the sternotomy and donor site wounds for the CABG patients

SUMMARY:
RCT on post-cardiac surgery patients using silver dressings vs. standard care. Conducted in ICU, CCU, telemetry units. Outcomes assessed via checklist & modified Parsonnet Score. Descriptive & inferential statistics for analysis.

DETAILED DESCRIPTION:
Background The prevalence of surgical site infections in cardiac surgery is about 10%. About 3% of patients who develop an SSI will die as a result. Multiple studies confirm that SSIs are complications with significant sequelae, such as longer hospitalization, increased health costs, increased morbidity, and mortality. Hence, the prevention and management of wound infections in median sternotomy incisions after adult cardiac surgery are crucial for optimizing patient outcomes, 5 Aim To assess the effect of the silver dressing on SSI rates in adult patients post-cardiac surgery.

Methodology A single-center randomized control trial approach will be employed. Adult patients admitted post-cardiac surgery with a sternotomy incision will be randomized into the intervention (n=78) or control group (n=77). Units will include the cardiac surgical intensive care unit, the coronary care unit, and the cardiovascular telemetry unit. The intervention will include the use of a silver dressing on the sternotomy incisions and the donor sites where applicable. The control group will follow standard care processes. Data collection will include a checklist and the modified Parsonnet Score. Data analysis will include descriptive and inferential statistics.

Conclusion The current rate of surgical site infection amongst cardiac surgical patients is 2.1 below the benchmark of 2.9 with an operational goal of 2.1.

ELIGIBILITY:
Inclusion Criteria:

Patients 18 years of age and older are scheduled for cardiac surgery requiring a sternotomy incision.

Exclusion criteria Presence of a concurrent infection and any systemic antibiotic other than those used for perioperative prophylaxis.

Patients who died without an infection within thirty days following surgery. Patients who had undergone another procedure through the same incision(s) within a year after enrollment in this study.

Patients who are a redo- such as needing debridement or an infection. Patients who have an open chest Patients on ECHMO Patients excessively bleeding Patients who require the surgery as an emergency Patients with a known allergy to silver dressings

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
silver dressing on SSI rates as compared to the standard dressing- Mepilex foam dressing in reducing SSIs. | 30 days post op

CONTACTS AND LOCATIONS:
Locations (1):
- King Faisal Specialist Hospital and Research Center - Jeddah, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
The data will not be shared due to privacy concerns and institutional policies.

REFERENCES:
- [Background] Dissemond J, Bottrich JG, Braunwarth H, Hilt J, Wilken P, Munter KC. Evidence for silver in wound care - meta-analysis of clinical studies from 2000-2015. J Dtsch Dermatol Ges. 2017 May;15(5):524-535. doi: 10.1111/ddg.13233. PMID 28485879

DOCUMENTS (1):
  • Study Protocol (2024-02-16): https://cdn.clinicaltrials.gov/large-docs/40/NCT07008040/Prot_000.pdf